CLINICAL TRIAL: NCT02360956
Title: Efficacy Study of Olmesartan Medoxomil on Coronary Atherosclerosis Progression and Epicardial Adipose Tissue(EAT) Volume Reduction in Patients With Coronary Atherosclerosis Detected by Coronary CT Angiography(CCTA)
Brief Title: Efficacy Study of Olmesartan Medoxomil on Coronary Atherosclerosis and Epicardial Adipose Tissue(EAT)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yundai Chen, Director of Cardiology,People's Liberation Army General Hospital, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2014-119-01
Record Dates: First submitted 2015-01-15; First posted 2015-02-11 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Coronary Atherosclerosis
Keywords: Olmesartan medoxomil; Epicardial adipose tissue; Multidetector Computed Tomography
MeSH Terms: conditions — Coronary Artery Disease | interventions — Olmesartan Medoxomil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olmesartan medoxomil (Experimental): Drug: Olmesartan medoxomil tablets(Daiichi Sankyo Inc, Japan). The initial dose is 20mg once daily. If blood pressure requiring further reduction after two weeks, olmesartan medoxomil may be increased to 40mg once daily.
  Interventions: Drug: Olmesartan medoxomil tablets
- Antihypertensive medication (Active Comparator): Drug:Any antihypertensive medication alone or in combination.Calcium channel blockers (CCBs),diuretics, beta-blockers, or other antihypertensive medication except angiotensin-Converting Enzyme Inhibitors inhibitors (ACEIs) or angiotensin II receptor blockers (ARBs).
  The drug dose must be individualized.
  Interventions: Drug: Antihypertensive medication (per doctor suggestion)

INTERVENTIONS:
Drug: Olmesartan medoxomil tablets — Dosage must be individualized. The usual recommended starting dose of Benicar is 20mg once daily when used as monotherapy in patients who are not volume-contracted.For patients requiring further reduction in blood pressure after 2 weeks of therapy, the dose of Benicar may be increased to 40 mg. Doses above 40 mg do not appear to have greater effect. Twice-daily dosing offers no advantage over the same total dose given once daily.
  Other Names: Benicar
  Arms: Olmesartan medoxomil
Drug: Antihypertensive medication (per doctor suggestion) — Any antihypertensive medication alone or in combination.Calcium channel blockers (CCBs),diuretics, beta-blockers, or other antihypertensive medication except ACE inhibitors or ARBs.The drug dose must be individualed.Dosage must be individualized.The patients should take the antihypertensive drugs according to doctors'suggestion.
  Other Names: no other names
  Arms: Antihypertensive medication

SUMMARY:
The purpose of this study is to determine whether olmesartan medoxomil is effective in the treatment of coronary atherosclerosis progression and epicardial adipose tissue(EAT) volume reduction in patients with coronary atherosclerosis detected by coronary CT angiography(CCTA).

DETAILED DESCRIPTION:
Epicardial adipose tissue(EAT) is directly deposited around the pericardium and coronary artery. By means of paracrine action, it can generate various kinds of cytokines, inflammatory factor and free fatty acids, that can affect the state of coronary endothelial function, inflammation and oxidative stress, which finally aggravate the progression of coronary atherosclerosis. In recent years, clinical studies have shown that EAT is a newly discovered independent risk factor of coronary atherosclerosis.Studies confirm that olmesartan medoxomil can improve endothelial function, resisting thrombosis, improve tissue reconstruction, resisting oxidative stress so as to achieve atherosclerosis resistant. Latest researches show that olmesartan medoxomil can better inhibit rat epididymal adipose cell hypertrophy and inflammatory reaction. Coronary CT angiography(CCTA) has emerged as a noninvasive imaging method for analysis coronary atherosclerosis. The purpose of this study is to determine whether olmesartan medoxomil is effective in the treatment of coronary atherosclerosis progression and EAT volume reduction in patients with coronary atherosclerosis detected by CCTA.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery stenosis between 30% and 70% determined by CCTA in essential hypertension patients
* resting diastolic blood pressure (DBP) between 90 and 110 mmHg
* type A and B for coronary artery vascular lesions

Exclusion Criteria:

* secondary hypertension
* coronary artery stenosis less than 30% or greater than 70% determined by CCTA
* contraindications to treatment with olmesartan medoxomil (allergy, glaucoma, digestive ulcer, is currently taking phosphodiesterase-5 inhibitor)
* resting systolic blood pressure (SBP) > 200 mmHg or resting diastolic blood pressure (DBP) > 110 mmHg
* Severe calcification, distortion or type C for coronary artery vascular lesions
* pregnancy
* unwillingness or inability to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Coronary atherosclerosis progression detected by CCTA | 12 month
  Coronary atherosclerosis progression is defined as ≥10% diameter reduction or progression of a pre-existing coronary stenosis; or ≥0.2mm reduction or progression of the minimal luminal area (MLD) in the lesion
Epicardial Adipose Tissue(EAT) volume detected by CCTA | 12 month

SECONDARY OUTCOMES:
The relationship between coronary atherosclerosis and EAT, as indicated by coronary atherosclerosis progression and epicardial adipose tissue(EAT) volume changes | 12 month
Serum levels of blood lipids | 12 month
  Blood lipids include total cholesterol,triglyceride,high density lipoprotein(HDL) and low density lipoprotein(LDL).
Serum levels of blood glucose | 12 month
  Blood glucose is defined as fasting blood glucose(FBG).
Circulating surrogate markers of atherosclerosis inflammation including hs-CRP,IL-6,MCP-1,TNF--α and MMP-9 | 12 month
  CRP: C reactive protein; IL: Interleukin; MCP: Monocyte chemotactic protein,composite of chemoattractant markers; TNF-α: tumor necrosis factor; MMP: Matrix metalloproteinase.
Individual circulating surrogate markers of endothelial function including NO and ET-1 | 12 month
  ET: Endothelin
Individual circulating surrogate markers of adipose tissue inflammation and metabolism including adiponectin and leptin. | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Chen Yundai, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

REFERENCES:
- [Background] Alexopoulos N, McLean DS, Janik M, Arepalli CD, Stillman AE, Raggi P. Epicardial adipose tissue and coronary artery plaque characteristics. Atherosclerosis. 2010 May;210(1):150-4. doi: 10.1016/j.atherosclerosis.2009.11.020. Epub 2009 Nov 20. PMID 20031133
- [Background] Cherian S, Lopaschuk GD, Carvalho E. Cellular cross-talk between epicardial adipose tissue and myocardium in relation to the pathogenesis of cardiovascular disease. Am J Physiol Endocrinol Metab. 2012 Oct 15;303(8):E937-49. doi: 10.1152/ajpendo.00061.2012. Epub 2012 Aug 14. PMID 22895783
- [Background] Ferrario C. Effect of angiotensin receptor blockade on endothelial function: focus on olmesartan medoxomil. Vasc Health Risk Manag. 2009;5(1):301-14. doi: 10.2147/vhrm.s3141. Epub 2009 Apr 8. PMID 19436655
- [Background] Maeda A, Tamura K, Wakui H, Ohsawa M, Azushima K, Uneda K, Kanaoka T, Kobayashi R, Ohki K, Matsuda M, Tsurumi-Ikeya Y, Yamashita A, Tokita Y, Umemura S. Effects of the Angiotensin receptor blocker olmesartan on adipocyte hypertrophy and function in mice with metabolic disorders. Biomed Res Int. 2014;2014:946492. doi: 10.1155/2014/946492. Epub 2014 Jun 2. PMID 24991574
- [Derived] Zhou Y, Tian F, Wang J, Yang JJ, Zhang T, Jing J, Chen YD. Efficacy study of olmesartan medoxomil on coronary atherosclerosis progression and epicardial adipose tissue volume reduction in patients with coronary atherosclerosis detected by coronary computed tomography angiography: study protocol for a randomized controlled trial. Trials. 2016 Jan 6;17:10. doi: 10.1186/s13063-015-1097-z. PMID 26739013